CLINICAL TRIAL: NCT04677322
Title: OBSERVATIONAL STUDY TO ASSESS THE EFFECTIVENESS OF THE INTERVENTION OF THE LOW-SODIUM DIET THROUGH THE MONITORING OF SODIUM IN URINE IN PATIENTS WITH HIGH BLOOD PRESSURE IN THE PRIMARY CARE SETTING
Brief Title: TO ASSESS THE EFFECTIVENESS OF THE INTERVENTION OF THE LOW-SODIUM DIET IN PATIENTS WITH HTA
Acronym: IDI-HTA2020
Status: Terminated | Type: Observational
Why Stopped: the principal investigator withdraws from the project for personal reasons
Sponsor: Instituto de Investigación Marqués de Valdecilla (Other)
Responsible Party: Sponsor
Other Study IDs: IDI-HTA-2020-01
Record Dates: First submitted 2020-12-09; First posted 2020-12-21 (Actual); Last update posted 2023-03-02 (Actual); Status verified 2023-02

CONDITIONS: Arterial Hypertension; Sodium Urine; Primary Care Center; Diet Habit
MeSH Terms: conditions — Hypertension; Feeding Behavior | interventions — Therapeutics

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Adult patients diagnosed and treated for high blood pressure — Educational program interventions conducted by primary care staff to encourage adherence to a low-sodium diet consisting of direct action on the patient and provision of educational materials will be assessed. Compliance and follow-up of the low sodium diet will be done by monitoring the sodium in urine in the target population, selected according to the selection criteria described in the protocol.

SUMMARY:
Arterial hypertension is an independent vascular risk factor and a frequent reason for consultation in Primary Care. It generates high cardiovascular morbidity and mortality (stroke, heart disease, kidney failure and other diseases). Moreover, given that it is a modifiable factor and that there are intervention and control measures that would lead to a significant reduction in cardiovascular incidence and morbimortality, it can be stated that ETS is a major public health problem.

The approach to this risk factor can be pharmacological and non-pharmacological. The non-pharmacological approach is based on lifestyle modification. Among the measures aimed at modifying lifestyles is the restriction of daily intake of sodium in the diet. Such restriction enhances the hypotensive effect of pharmacological treatment so that its application and intensification would delay the start of pharmacological therapy, as well as avoid the need to increase the dose of antihypertensive drugs or the number of drugs to be used for the control of hypertension.

In relation to salt intake in the Spanish population, the average is above the figures of less than 5 grams per day recommended by the WHO. Sodium intake can be estimated by determining the 24-hour urine sodium concentration. In addition, there is a positive correlation between systolic and diastolic blood pressure figures and the excretion of sodium in urine.

DETAILED DESCRIPTION:
In the present work, with a prospective cohort observational study design, it intends to assess the effectiveness of the use of an educational program based on the follow up of a hyposodium diet and assessed through the routine use of urine sodium monitoring of the hypertensive patient in the primary care setting, in order to optimize treatment, as well as to review the clinical control in this group of patients. On the other hand, it is intended to establish guidelines in the form of practical guidelines to provide with a standardized clinical approach for primary care centers.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 40 years old.
* Patients diagnosed with HTA (according to criteria ESC/ESH 2018) in a PA consultation or through MAP at the health center.
* In treatment with single, double or triple antihypertensive therapy.
* Patients with ST figures ≥140.
* Patients with TD numbers ≥90.
* Patients with stable antihypertensive treatment or without modifications in the treatment at least in the last month.
* Patients who commit to follow up the study.
* Patients who have given written informed consent.

Exclusion Criteria:

* Patients with decompensated heart failure
* Severe renal failure.
* Decompensated liver disease.
* Taking non-insulin antidiabetic
* Hypertension of pharmacological origin and other causes.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed and treated for high blood pressure
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2022-09-01 (Actual)

PRIMARY OUTCOMES:
Systolic and diastolic TA values, the upper limit being 140 (systolic) and the lower range 90 (diastolic). | basal
Systolic and diastolic TA values, the upper limit being 140 (systolic) and the lower range 90 (diastolic). | 6 months

SECONDARY OUTCOMES:
Sodium and potassium levels in 24-hour urine and isolated urine sample, with sodium limits of 20 mEq/L in a random urine sample and 40 to 220 mEq per day. | basal
Sodium and potassium levels in 24-hour urine and isolated urine sample, with sodium limits of 20 mEq/L in a random urine sample and 40 to 220 mEq per day, after educational intervention. | 6 months
To analyze the use of antihypertensive drugs USING morisk-green test, after educational intervention | 6 months
To verify compliance with the hyposodium diet and pharmacological treatment through the use of EuroQol-5D questionnaires | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Centro de salud Astillero, Santander, Cantabria, Spain